CLINICAL TRIAL: NCT04063449
Title: A Controlled Clinical Study of Endostar/PD-1 Inhibitors Combined With PP as First-line Treatment for Advanced Non-squamous Cell Lung Cancer With Negative Driving Gene
Brief Title: Endostar/PD-1 Inhibitors Combined With PP for Advanced NSCLC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dong Wang (Other)
Responsible Party: Sponsor-Investigator, Dong Wang, chief physician, Third Military Medical University
Organization: Third Military Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ThirdMMU09
Record Dates: First submitted 2019-08-19; First posted 2019-08-21 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Non-squamous Non-small Cell Lung Cancer
Keywords: Non-squamous NSCLC；endostar;PD-1 inhibitor;chemotherapy
MeSH Terms: interventions — endostar protein

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental:group A (Experimental): endostar,210 mg,CIV 72h,d1-d3; sintilimab,200mg,IV,d1; carboplatin,5/AUC,IV,d1; Pemetrexed,500mg/m2 ,IV,d1； 3 weeks for a cycle;4-6 cycles; after the treatment for 4-6 cycles,endostar plus sintilimab for maintenance therapy until PD or intolerable toxicity ;
  Interventions: Drug: endostar/PD-1 inhibitor
- control:group B (Active Comparator): endostar,210 mg,CIV 72h,d1-d3; carboplatin,5/AUC,IV,d1; Pemetrexed,500mg/m2 ,IV,d1； 3 weeks for a cycle;4-6 cycles; after the treatment for 4-6 cycles,endostar for maintenance therapy until PD or intolerable toxicity ;
  Interventions: Drug: endostar

INTERVENTIONS:
Drug: endostar/PD-1 inhibitor — Antiangiogenic therapy plus immunotherapy and chemotherapy
  Arms: Experimental:group A
Drug: endostar — Antiangiogenic therapy plus chemotherapy
  Arms: control:group B

SUMMARY:
A Controlled Clinical Study of Endostar/PD-1 Inhibitors Combined With chemotherapy(Carboplatin-Pemetrexed) as First-line Treatment for Advanced Non-squamous Cell Lung Cancer With Negative Driving Gene

DETAILED DESCRIPTION:
This study was a controlled clinical trial.A total of 170 patients with pathologically confirmed non-squamous NSCLC would be enrolled.Patients were randomly divided into two groups, with 85 in the group A and 85 in the group B.The group A was treated with endostar,sintilimab and chemotherapy(carboplatin-pemetrexed).The group B was treated with endostar and chemotherapy(carboplatin-pemetrexed).The efficacy and safety would be evaluated.The progression-free survival and overall survival would be analyzed.This data of this study might provide a more effective treatment for non-squamous NSCLC.

ELIGIBILITY:
Inclusion Criteria:

1. Patients volunteered to participate in the study and signed the informed consent;
2. Age 18-75, both male and female;
3. Histologically or cytologically confirmed advanced or metastatic (stage III B, III C or IV) non-squamous NSCLC , and no mutation was detected in the driving gene.
4. At least one measurable lesion according to RECIST 1.1,which should not be treated locally, such as radiotherapy.
5. ECOG PS 0-1
6. Expected survival ≥ 3 months
7. Patients who never received systemic therapy in the past, including radiotherapy ,chemotherapy, targeted therapy and immunotherapy , or patients who relapsed more than 6 months after adjuvant chemotherapy.
8. The main organ functions accorded with the following criteria within 7 days before treatment:

(1)Blood routine examination ( without blood transfusion in 14 days): hemoglobin (HB) ≥ 90 g/L; neutrophil absolute value (ANC) ≥ 1.5 *109/L; platelet (PLT) ≥80 *109/L.

(2) Biochemical tests should meet the following criteria: 1) total bilirubin (TBIL) ≤1.5 times of upper limit of normal (ULN); 2) alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 *ULN, if accompanied by liver metastasis, ALT and AST ≤ 5* ULN; 3) serum creatinine (Cr) ≤ 1.5* ULN or creatinine clearance rate (CCr) ≥ 60 ml/min;4) Serum albumin (≥35g/L).

(3) Doppler echocardiography: left ventricular ejection fraction (LVEF) ≥the low limit of normal value (50%).

9 Tissue samples should be provided for biomarker analysis (such as PD-L1 ) Patients who could not provide new tissues could provide 5-8 paraffin sections of 3-5 μm by archival preservation.

Exclusion Criteria:

1. Severe allergic reactions to humanized antibodies or fusion proteins in the past
2. known to have hypersensitivity to any component contained in Endostar or antibody preparations;
3. Diagnosed of immunodeficiency or received systemic glucocorticoid therapy or any other form of immunosuppressive therapy within 14 days before the study, allowing physiological doses of glucocorticoids (≤10 mg/day prednisone or equivalent);
4. Patients with active, known or suspected autoimmune diseases. Patients with type I diabetes, hypothyroidism requiring hormone replacement therapy, skin disorders requiring no systemic treatment (such as vitiligo, psoriasis or alopecia). Patients who would not triggers can be included.
5. Serious heart disease, include congestive heart failure, uncontrollable high-risk arrhythmia, unstable angina pectoris, myocardial infarction, and severe valvular disease.
6. Patients treated targeted drugs such as bevacizumab, sunitinib, sorafenib, imatinib, famitinib, regiffenil, apatinib and anlotinib
7. Patients recieved systemic antineoplastic therapy, including cytotoxic therapy, signal transduction inhibitors, immunotherapy (or mitomycin C within 6 weeks before the grouping),recieved over-extended-field radiotherapy (EF-RT) within 4 weeks before the grouping or limited-field radiotherapy to evaluate the tumor lesions within 2 weeks before the grouping
8. Positive hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus antibody (HCV Ab), indicating acute or chronic infection.
9. Patients with active pulmonary tuberculosis (TB) infection judged by chest X-ray examination, sputum examination and clinical physical examination. Patients with active pulmonary tuberculosis infection in the previous year should be excluded even if they have been treated; Patients with active pulmonary tuberculosis infection more than a year ago should also be excluded unless the course and type of antituberculosis treatment previously were appropriate.
10. Patients with brain metastases with symptoms or symptoms controlling less than 2 months
11. Major surgical treatment, incision biopsy or significant traumatic injury were performed within 28 days before the grouping.
12. The imaging showed that the tumors had invaded important blood vessels or likely to invade important blood vessels and cause fatal massive hemorrhage during the follow-up period judged by researchers.
13. patients with any physical signs or history of bleeding; Patients with any bleeding or bleeding events ≥ CTCAE grade 3,unhealed wounds, ulcers or fractures within 4 weeks before grouping
14. Arteriovenous thrombosis occurred within 6 months, such as cerebrovascular accident (including temporary ischemic attack), deep vein thrombosis and pulmonary embolism.
15. The study is dangerous for patients judged by researcher, or patients who may affect the completion of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2019-08-20 (Estimated); Primary Completion 2020-06-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
progression-free survival(PFS) | approximately 36 months
  progression-free survival is defined as the time from enrollment to the date of first document disease progression or death from any cause
overall survival (OS) | approximately 36 months
  overall survival is defined as the time from randomization to death from any cause

SECONDARY OUTCOMES:
objective response rate(ORR) | approximately 18 months
  complete response(CR)+partial response(PR) according to RECIST 1.1
adverse event(AE) | approximately 36 months
  adverse event according to NCI CTCAE V4.0

CONTACTS AND LOCATIONS:
Overall Officials: Dong Wang, PH.D, Principal Investigator — Daping Hospital, Third Military Medical University, Chongqing,China
Locations (1):
- Daping Hospital, Third Military Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided